CLINICAL TRIAL: NCT05633888
Title: Prospective, Multi-Center, Single Arm Post-Market Feasibility Study of the Tenon Medical CATAMARAN™ SI Joint Fusion System
Brief Title: Post-Market Feasibility Study of the Tenon Medical CATAMARAN™ SI Joint Fusion System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tenon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL015
Record Dates: First submitted 2022-11-14; First posted 2022-12-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sacroiliac Joint Disruption; Degenerative Sacroiliitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CATAMARAN SI Joint Fusion System (Experimental): Placement of the Catamaran Fixation Device
  Interventions: Device: CATAMARAN SI Joint Fusion System

INTERVENTIONS:
Device: CATAMARAN SI Joint Fusion System — Placement of the Catamaran Fixation Device

SUMMARY:
The purpose of this study is to evaluate the outcomes of patients with sacroiliac joint pain treated with the CATAMARAN SI Joint Fusion System.

DETAILED DESCRIPTION:
This is a multi-center post-market study to evaluate the clinical outcomes of patients with sacroiliac joint disruptions or degenerative sacroiliitis treated with the CATAMARAN SI Joint Fusion System.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sacroiliac joint disruption or degenerative sacroiliitis based on ALL of the following:

  * Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test), and
  * Patient has at least 3 of 5 physical examination maneuvers specific for SI joint pain (Fabers, Compression, Distraction,Thigh thrust, Gaenslen's test, and/or Sacral thrust test), and
  * Patient has improvement in lower back pain VAS of at least 50% of the pre injection VAS after fluoroscopic controlled injection of local anesthetic into affected SI joint(s) (including previous documented test <6 months ago)
* Patient has failed conservative care (non-surgical) > 6 months
* Patient has a pre-operative Oswestry Disability Index score > 30%
* Patient has a pre-operative SI joint pain score of > 50 on a 0-100 mm visual analog scale (VAS)
* Patient, or authorized representative, signs a written Informed Consent form to participate in the study
* Patient is willing and able to complete study follow-up requirements

Exclusion Criteria:

* Planned bi-lateral SI joint fixation
* Severe lower back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, and lumbar vertebral body fracture (this is done by physical exam, medical history, and MRI/CT/X-ray as required)
* Other known sacroiliac pathology such as: sacral dysplasia, inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA- associated spondyloarthropathy), tumor, acute fracture, crystal arthropathy
* History of recent (<1 year) fracture of the pelvis with documented malunion, non-union of sacrum or ilium or any type of internal fixation of the pelvic ring
* Severe osteoporosis
* Paget's disease, osteomalacia, osteomalacia or other metabolic bone disease
* Any condition or anatomy that makes treatment with the CATAMARAN SI Joint Fusion System infeasible including deformity
* Known allergy to titanium or titanium alloys
* Morbid obesity
* Active malignancy: a history of any invasive malignancy (except non-melanoma skin cancer), unless the subject has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least five years
* Patient has systemic infection or active infection at the treatment site
* Chronic rheumatologic condition (e.g., rheumatoid arthritis)
* Patient has uncontrolled diabetes
* Patient is currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation
* Prominent neurologic condition that would interfere with physical therapy
* Patient is pregnant or wishes to become pregnant in the next two years
* Patient is not likely to comply with the follow-up evaluation schedule
* Patient is participating in a clinical trial of another investigational drug or device in which the primary endpoint has not occurred
* Patient has a psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation
* Known or suspected drug or alcohol abuse
* Patient is a prisoner or a ward of the state

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects that meet the definition of Subject Success at 6 months post-procedure | 6 months post procedure
  Change from baseline in VAS SI joint pain score to be reduced by at least 20 mm, Lack of device-related serious adverse events, Absence of neurologic worsening related to the sacral spine compared to baseline (unless attributable to a concurrent medical condition or other cause unrelated to the device and/ or study procedure), and Absence of surgical re-intervention (removal, revision, reoperation, or supplemental fixation) for SI joint pain.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Northwest Specialty Hospital, Coeur d'Alene, Idaho
  - Comprehensive Pain and Spine Specialists, Muncie, Indiana
  - Vitality Pain Centers, Louisville, Kentucky
  - Orthopedic Associates of Duluth, Duluth, Minnesota
  - St. Louis Pain Consultants, Chesterfield, Missouri
  - St. George Orthopedic Spine, St. George, Utah

IPD SHARING:
Plan to Share IPD: No